CLINICAL TRIAL: NCT03277508
Title: Assistive Soft Robotic Glove Intervention Using Brain-Computer Interface for Elderly Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other); Agency for Science, Technology and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 2017/00312
Record Dates: First submitted 2017-04-21; First posted 2017-09-11 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Stroke
Keywords: Brain-computer integration
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A randomization stratification method, with a computer generated random sequence will be used. Subjects will be grouped in strata according to their Fugl-Meyer scores(0-28 vs 29-45) and randomized separately according to a block randomization to receive either of following treatments:(1) Treatment A: 18 sessions for 6 weeks of 60 minutes of passive robot-assisted hand therapy+ 30 minutes of standard hand therapy.(2) Treatment B: 18 sessions for 6 weeks of 60 minutes of BCI controlled robot-assisted hand therapy + 30 minutes of standard hand therapy.
Who Masked: Outcomes Assessor
Masking Description: The blinding will be carried out in such a way that the therapist will provide conventional therapy and assess the arm function without knowing the group that the patients belong to. The BCI Robot and Passive Robot will be administered by other study team member. A third party study team member not participating in the intervention will keep the log book which contains information regarding patients study ID and group. Randomization codes will be broken when all interventional and follow-up sessions were completed or when the patient decides to quit participation. The third party team member will unmask according to PI's request in this occasion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCI robot assisted hand therapy (Experimental): Brain-computer integration robot assisted hand therapy
  Interventions: Device: BCI Robot Assisted Hand Therapy
- CPM robot assisted hand therapy (Active Comparator): Continue Passive Movement robot assisted hand therapy
  Interventions: Device: CPM Robot Assisted Hand Therapy

INTERVENTIONS:
Device: BCI Robot Assisted Hand Therapy — 18 sessions (3 times per week for a total of 6 weeks) of 1.5 hours each training (60 minutes of BCI Robot and 30 minutes of the standard hand therapy).
  Session 1-3. Peg game: Lateral movement of gears/cups Session 4-6. Moving cups onto a shelf: Elevation process for the arm, small cups to be used.
  Session 7-9. Carrying of basket: Heavier load to be used, patient to hold the basket by the handles at the side, not by its base.
  Session 10-12. Opening bottle + pouring into a cup: Training of ADL Session 13-15. Eating: Use of a modified spoon to train ADL Session 16-18. Box and blocks: Precise index finger and thumb control
  Arms: BCI robot assisted hand therapy
Device: CPM Robot Assisted Hand Therapy — 18 sessions (3 times per week for a total of 6 weeks) of 1.5 hours each training (60 minutes of Passive Robot and 30 minutes of the standard hand therapy).The procedure will include the following: Session 1-18: Continuous passive motion
  Arms: CPM robot assisted hand therapy

SUMMARY:
This research aims to integrate and develop a novel Brain-Computer Interface (BCI) controlled soft robotic glove, evaluate the ability of the glove in achieving common hand grasping postures and to assess the efficacy of the glove in assisting stroke patients with completing functional tasks. The BCI-controlled soft robotic glove utilizes patients' user intent to deliver specific electroencephalographic patterns that can trigger robot-assisted hand movement to the affected hand.

DETAILED DESCRIPTION:
Hand motor impairment is very common after a stroke. These impairments include difficulty moving and coordinating the hands and fingers, which inhibits stroke patients from being able to perform daily functional tasks independently, resulting in a reduced quality of life. More than half of people with upper limb impairment after stroke will still have problems many months to years after their stroke. Therefore, improving hand function is a core element of rehabilitation. Many possible interventions have been developed; these may involve different exercises or training, specialist equipment or techniques, or they could take the form of a drug (pill or injection) given to help hand movement. There is limited evidence that suggests the following interventions may be effective: constraint-induced movement therapy, mental practice, mirror therapy,interventions for sensory impairment, virtual reality and a relatively high dose of repetitive task practice. Current hand rehabilitation robotic devices are typically driven by rigid linkages or joints, which subject the patient's fingers into a single plane of motion that will feel unnatural and uncomfortable. On top of that,these devices belong to the class of continuous passive motion (CPM) devices that only promote hand range-of-motion, but do not require the patient to play a semi-active role in performing the hand exercises. Furthermore, there is a huge demand for solutions assisting stroke patients with using the densely paralyzed hand to perform activities of daily living (ADL) in real life, which is not available at present. Most of the hand rehabilitation robotic devices available in the market cannot assist paralyzed hand to carry out ADL. To develop an assistive device to solve this unmet need, we decided to combine BCI technology with the wearable soft robotic glove, which enables actuation of paralyzed hand by motor imagery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55-90 years regardless of lesion size, race
* History of stroke less than 3 months prior to participation
* Stroke type: ischemic or haemorrhagic
* Fugl-Meyer motor score (FM score) of upper extremity impairment of 0-45 out of a maximum score of 66 on the Fugl-Meyer assessment scale
* Ability to pay attention and maintain supported sitting for 1.5 hours continuously
* Lack of or poor hand mobility (Medical Research Council Grade ≤ 2/5)
* Able to give own consent
* Able to comprehend and follow commands (Abbreviated Mental Test equal or more than 7)
* Fulfil BCI resting brain states on initial screening.
* Unilateral upper limb impairment

Exclusion Criteria:

* Recurrent clinical stroke
* Functional status: severe aphasia or inattention, unstable medical conditions which may affect participation (e.g. unresolved sepsis, postural hypotension) or anticipated life expectancy of <1 year due to malignancy or neurodegenerative disorder)
* Hemispatial neglect (visual or sensory) or severe visual impairment despite visual aids
* History of severe depression or active psychiatric disorder
* Skull defect or previous cranial surgery as this would affect physical fit of EEG cap interface
* Local arm factors: severe spasticity Modified Ashworth scale >1+ in any region, fixed joint contractures or joint replacements, patients with poor skin conditions which would contraindicate repetitive arm training, upper limb pain impeding movements with visual analogue scale (VAS score) >4/10, other conditions ensuing upper limb weakness, skull defect, polydactyly or amputation of fingers, and allergy to electrodes or adhesive gel

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test | 30 minutes
  It assesses a client's ability to handle objects differing in size, weight and shape and therefore can be considered to be an arm-specific measure of activity limitation
Fugl-Meyer Assessment | 20 minutes
  It is designed to assess motor functioning, balance, sensation and joint functioning.
Grip Strength Test | 5 minutes
  The purpose of this test is to measure the maximum isometric strength of the hand and forearm muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hoon Lim, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] F.Z. Low, H.K. Yap, J.H. Lim, F. Nasrallah, J.C.H. Goh, C.H. Yeow. Wearable Soft Robotics for Rehabilitation. 8th Asian Pacific Conference on Biomechanics 2015 (Sapporo).
- [Background] H.K. Yap, F. Nasrahllah, J.H. Lim, F.Z. Low, J.C.H. Goh, C.H. Yeow. MRC-Glove: A fMRI Compatible Soft Robotic Glove for Hand Rehabilitation Application, 14th IEEE/RAS-EMBS International Conference on Rehabilitation Robotics (ICORR 2015).
- [Background] H.K. Yap, J.H. Lim, F. Nasrahllah, J.C.H. Goh, C.H. Yeow. A Soft Exoskeleton for Hand Assistive and Rehabilitation Application Page 8 using Pneumatic Actuators with Variable Stiffness, in IEEE Int. Conf. Robotics and Automation 2015.
- [Background] H.K. Yap, J.C.H. Goh, C.H. Yeow. Design and Characterization of Soft Actuator for Hand Rehabilitation Application. 6th European Conference of the International Federation for Medical and Biological Engineering (MBEC 2014)
- [Background] H.K. Yap, J.H. Lim, F. Nasrallah, J.C.H. Goh, C.H. Yeow. Customizable Pneumatic Bending Actuator for Finger Rehabilitation. Design of Medical Devices Conference Europe 2014 (Delft)
- [Background] C.H. Yeow, A.T. Baisch, S.G. Talbot, C.J. Walsh. Differential spring stiffness design for finger therapy exercise device: bio-inspired from stiff pathological finger joints. ASME Journal of Medical Devices 2012
- [Background] Ang KK, Chin ZY, Wang C, Guan C, Zhang H. Filter Bank Common Spatial Pattern Algorithm on BCI Competition IV Datasets 2a and 2b. Front Neurosci. 2012 Mar 29;6:39. doi: 10.3389/fnins.2012.00039. eCollection 2012. PMID 22479236
- [Background] Ang KK, Guan C, Phua KS, Wang C, Zhao L, Teo WP, Chen C, Ng YS, Chew E. Facilitating effects of transcranial direct current stimulation on motor imagery brain-computer interface with robotic feedback for stroke rehabilitation. Arch Phys Med Rehabil. 2015 Mar;96(3 Suppl):S79-87. doi: 10.1016/j.apmr.2014.08.008. PMID 25721551
- [Background] Ang KK, Chua KS, Phua KS, Wang C, Chin ZY, Kuah CW, Low W, Guan C. A Randomized Controlled Trial of EEG-Based Motor Imagery Brain-Computer Interface Robotic Rehabilitation for Stroke. Clin EEG Neurosci. 2015 Oct;46(4):310-20. doi: 10.1177/1550059414522229. Epub 2014 Apr 21. PMID 24756025
- [Background] Ang KK, Guan C, Phua KS, Wang C, Zhou L, Tang KY, Ephraim Joseph GJ, Kuah CW, Chua KS. Brain-computer interface-based robotic end effector system for wrist and hand rehabilitation: results of a three-armed randomized controlled trial for chronic stroke. Front Neuroeng. 2014 Jul 29;7:30. doi: 10.3389/fneng.2014.00030. eCollection 2014. PMID 25120465
- [Background] Rojas JI, Zurru MC, Romano M, Patrucco L, Cristiano E. Acute ischemic stroke and transient ischemic attack in the very old--risk factor profile and stroke subtype between patients older than 80 years and patients aged less than 80 years. Eur J Neurol. 2007 Aug;14(8):895-9. doi: 10.1111/j.1468-1331.2007.01841.x. PMID 17662011
- [Background] Rosamond W, Flegal K, Furie K, Go A, Greenlund K, Haase N, Hailpern SM, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell C, Roger V, Sorlie P, Steinberger J, Thom T, Wilson M, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2008 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2008 Jan 29;117(4):e25-146. doi: 10.1161/CIRCULATIONAHA.107.187998. Epub 2007 Dec 17. No abstract available. PMID 18086926
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Venketasubramanian N, Chen CL. Burden of stroke in Singapore. Int J Stroke. 2008 Feb;3(1):51-4. doi: 10.1111/j.1747-4949.2008.00181.x. PMID 18705915
- [Result] Hong Kai Yap, Kamaldin N, Jeong Hoon Lim, Nasrallah FA, Goh JCH, Chen-Hua Yeow. A Magnetic Resonance Compatible Soft Wearable Robotic Glove for Hand Rehabilitation and Brain Imaging. IEEE Trans Neural Syst Rehabil Eng. 2017 Jun;25(6):782-793. doi: 10.1109/TNSRE.2016.2602941. Epub 2016 Aug 25. PMID 28113591